CLINICAL TRIAL: NCT03303846
Title: Combined Breast MRI/Biomarker Strategies to Identify Aggressive Biology
Brief Title: Combined Breast MRI and Biomarker Strategies in Identifying High-risk Breast Cancer Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 17009; NCI-2017-01757 (Registry Identifier: NCI CTRP); U01CA189283 (NIH)
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Healthy Subject
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (breast MRI, biopsy) (Experimental): Participants undergo standard of care high risk breast cancer screening MRIs at baseline and follow-up and blood sample collection at baseline. Participants also undergo collection of breast tissue samples at any breast biopsy or breast surgery.
  Interventions: Procedure: Magnetic Resonance Imaging; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo high risk breast cancer screening MRI
  Other Names: Magnetic Resonance / Nuclear Magnetic Resonance; MRI; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial studies normal breast tissue changes combined with breast magnetic resonance imaging (MRI) that may suggest the beginnings of cancer development. Using breast tissue markers in combination with breast imaging such as MRI may help to more accurately assess a woman's risk of developing breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the number of high risk women with abnormal screening breast MRI and morphologically normal biopsy over 7 years.

SECONDARY OBJECTIVES:

I. To determine if WNT10B/mutant p53 expression as measured in the 0-month biopsy predicts women with an abnormal MRI/non-cancerous biopsy who will progress to cancer over 7 years.

TERTIARY OBJECTIVES:

I. To determine the predictive accuracy of WNT10B with MRI, of which will be compared with MRI alone using the C-index.

OUTLINE:

Participants undergo standard of care high risk breast cancer screening MRIs at baseline and follow-up and blood sample collection at baseline. Participants undergo collection of breast tissue samples at any breast biopsy or breast surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women who are undergoing screening breast MRI as per standard of care for high-risk breast cancer screening
* Willing to donate left-over tissue if patient undergoes a breast biopsy and/or breast surgery
* Willing to have about 40 mL of blood (approximately 3 tablespoons) drawn
* Documented informed consent of the participant

Exclusion Criteria:

* Allergy or intolerance to gadolinium
* Inability to undergo breast MRI (e.g. claustrophobia)
* Participants with active cancer diagnosis (exception: skin cancer, biopsy-proven atypical lobular, ductal hyperplasia and/or lobular carcinoma in situ)
* Previous diagnosis of stage 4 cancer
* Participants who have received cytotoxic chemotherapy within 1 year prior to screening breast MRI
* Participants who have received endocrine therapy within 1 year prior to screening breast MRI
* Participants who have received breast radiation within 1 year prior to screening breast MRI
* Radiation to both breasts
* Pregnant and/or lactating within 1 year prior to screening breast MRI
* Receives screening breast MRIs at an outside facility other than the consenting institution

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2026-04-25 (Estimated); Study Completion 2026-04-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of triple-negative breast cancer (invasive and/or ductal carcinoma in situ [DCIS]) within the 12-month period of the study | Up to 12 months
  Development of breast cancers other than triple-negative (e.g. estrogen receptor (ER), progesterone receptor (PR), human epidermal growth factor receptor 2 (HER2) the study analysis, however they will be reported as descriptive statistics.

SECONDARY OUTCOMES:
Expression of WNT10B/mutant p53 in morphologically normal breast tissue | Up to 12 months
  Biopsy tissue will be assessed for 1) activated WNT10B (measured by presence of high phospho-beta-catenin; present vs. absent) and 2) loss of p53 function (measured by the loss of p21 expression; present versus [vs.] absent). The optimal cut for the WNT10B to differentiate progression vs. non-progression women will be carried out by receiver operating characteristic (ROC) analysis, and hence WNT10B expression will be dichotomized to high vs. low expression. Chi-square test 12-month progression. Adjusted association will be further explored by logistic regression incorporating subject characteristics, such as age, body mass index (BMI), race, and BRCA1.

OTHER OUTCOMES:
Predictive accuracy of WNT10B with magnetic resonance imaging (MRI) | Up to 12 months
  The specificity for MRI combined with WNT10B and/or p53 based biomarkers to detect triple negative breast cancer (TNBC) will be calculated with 95% confidence interval (CI). Its prediction accuracy will be described by C-index and compared to that by diagnosis by MRI alone.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Seewaldt, MD, Principal Investigator — City of Hope Medical Center
Locations (5):
- United States (5):
  - City of Hope Medical Center, Duarte, California
  - University of Southern California, Los Angeles, California
  - Duke University, Durham, North Carolina
  - Ohio State University, Stefanie Spielman Comprehensive Breast Center, Columbus, Ohio
  - University of Wisconsin, Madison, Wisconsin